CLINICAL TRIAL: NCT04294277
Title: Open-label, Single-arm, Phase II Study, Evaluating Safety and Efficacy of INCB054828 (Pemigatinib) as Adjuvant Therapy for Molecularly-selected, High-risk Patients With Urothelial Carcinoma Who Have Received Radical Surgery
Brief Title: Safety and Efficacy of Pemigatinib in Patients With High-risk Urothelial Cancer After Radical Surgery
Acronym: PEGASUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Screening success and patient recruitment was much lower than projected and a clinical/scientific interpretation will not be possible.
Sponsor: European Association of Urology Research Foundation (Other)
Collaborators: Incyte Biosciences International Sàrl (Industry); AMS Advanced Medical Services GmbH (Industry); High Research s.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EAU RF 2018-02
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Results first posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Urothelial Cancer
Keywords: Urothelial carcinoma; FGFR inhibitor; Pemigatinib
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pemigatinib

STUDY DESIGN:
Intervention Model Description: Open-label, single-arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Treatment with Pemigatinib at the protocol-defined dose administered orally once daily as continuous therapy schedule until 12 months.
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — At Day 1, prior to the start of treatment, results from screening visit evaluations are reviewed to determine eligibility requirements. Subsequent visits during treatment phase will take place at Day 8, Day 15 and Day 21 and subsequently at 3 week intervals. Timing of subsequent visits can be prolonged to max. 9 week intervals if no problems exist during the first 12 weeks of therapy. Subjects will self-administer study drug using an oral QD regimen in a continuous dosing schedule. Each dose of Pemigatinib should be taken first thing in the morning upon waking or after a 2-hour fast; subjects should then fast for an additional 1 hour after taking study drug. The starting dose is 13.5 mg Pemigatinib. Study treatment will continue until 12 months, or until the evidence of disease relapse or onset of unacceptable toxicity.
  Other Names: INCB054828

SUMMARY:
The purpose of this clinical trial is to demonstrate the benefit of Pemigatinib, a drug that has indicated promising effects for relapse free survival in molecularly-selected, high-risk patients with urothelial carcinoma (UC) who have received radical surgery. Patients will receive Pemigatinib at a once-daily dose on a continuous schedule, continued until 12 months.

DETAILED DESCRIPTION:
This is an open-label, single-arm, Phase II study, evaluating safety and efficacy of INCB054828 (Pemigatinib) as adjuvant therapy for molecularly-selected, high-risk patients with urothelial carcinoma (UC) who have received radical surgery. Patients will receive Pemigatinib at a once-daily (QD) dose of 13.5 mg on a continuous schedule. Treatment will be continued until 12 months, or until the evidence of disease relapse or onset of unacceptable toxicity.

Hyperphosphatemia can be managed with diet modification, phosphate binders, or dose modification. Since mineralization of the cornea and retinal changes consisting of serous retinal detachment have been reported in humans, ophthalmic exams are done at baseline and once every 12 weeks during treatment and should include a visual acuity test, slit-lamp examination and fundoscopy. Additional assessments (e.g. Orbital computerized tomography (CT) should be done if clinically relevant retinal findings are observed on ophthalmologic exams and in participants with reported visual adverse events (AEs) or change in visual acuity, if the events or changes are suspected to be of retinal origin.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of pT3-4 and/or pN1-3 UC of the urinary bladder or upper urinary tract after radical cystectomy / radical nephroureterectomy. Patients with mixed histologies are required to have a dominant (i.e. at least 50%) urothelial cell carcinoma pattern.
* Previous administration of at least 3 cycles of neoadjuvant cisplatin-based chemotherapy OR, if neoadjuvant chemotherapy was not administered, ineligibility to receive cisplatin-based adjuvant chemotherapy based on Galsky's criteria, that include at least one of the following: (1) WHO performance status ≥ 2 and/or (2) creatinine-clearance < 60 ml/min and/or (3) CTCAE Gr ≥ 2 hearing loss and/or (4) CTCAE Gr ≥ 2 neuropathy.
* Evidence of FGFR alterations (mutations or translocations as specified in protocol) as assessed by a centralized Foundation Medicine test (Foundation One).
* Recovered with no evidence of disease confirmed by radiological images, prior to start of adjuvant therapy within 13 weeks after radical surgery.
* Willingness to avoid pregnancy or fathering children
* Written informed consent.

Exclusion Criteria:

* Any previous receipt of a selective FGFR inhibitor.
* Presence of primary CIS only.
* Presence of another malignancy in the 3 years before enrolment except for basal cell carcinoma or squamous cell carcinoma of the skin, cis of cervix, localised prostate cancer in active surveillance or other non invasive or other indolent malignancy that has undergone potentially curative therapy.
* Presence of pregnancy or lactation.
* Distant metastases (M1 disease).
* Treatment with other investigational drugs, receipt of anticancer medications (except for neoadjuvant cisplatin-based chemotherapy, see second inclusion criterion) or radiotherapy after radical surgery.
* Use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half lives (whichever is longer) before the first dose of study treatment.
* Abnormal laboratory parameters:

  * Total bilirubin ≥ 1.5 × upper limit of normal (ULN; ≥ 2.5 × ULN if Gilbert syndrome).
  * AST and/or ALT > 2.5 × ULN
  * Creatinine clearance ≤ 30 mL/min based on Cockroft-Gault.
  * Serum phosphate > institutional ULN.
  * Serum calcium outside of the institutional normal range or serum albumin-corrected calcium outside of the institutional normal range when serum albumin is outside of the institutional normal range.
* History of human immunodeficiency virus infection or active tuberculosis infection.
* Diagnosis of immunodeficiency or receiving chronic systemic steroid therapy (exceeding > 10 mg daily of prednison equivalent; inhalation steroids are permitted).
* Evidence of hepatitis B virus or hepatitis C virus active infection or risk of reactivation.
* Severe hepatic impairment
* Known prior severe hypersensitivity to investigational products or its excipients
* History of clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months of enrolment, New York Heart Association Class III or IV.
* Current evidence of corneal disorder/keratopathy (including but not limited to bullous/band keratopathy, corneal abrasion, inflammation/ulceration, keratoconjunctivitis, etc) or retinal disorder (including but not limited to, central serous retinopathy, macular/retinal degeneration, diabetic retino-pathy, retinal detachment, etc) as confirmed by ophthalmologic examination.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Necchi, Dr., Principal Investigator — IRCCS San Raffaele Hospital
Locations (5):
- Italy (5):
  - ASST Papa Giovanni XXIII, Bergamo
  - Policlinico Sant'Orsola-Malpighi - Azienda Ospedaliero-Univeristaria di Bologna, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IRCCS San Raffaele Hospital, Milan
  - Fondazione Policlinico Universitario A. Gemelli, IRCCS, Roma

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In 2020, the study was started in 5 Italian centers and recruitment commenced. The first patient was screened in July 2020.
Period: Overall Study
Arm/Group | Treatment Arm
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 73.5 [71 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Relapse-free Survival (RFS) After Start of Treatment With Pemigatinib.
Description: In the protocol, RFS at Year 2 was defined as the time from the start of treatment until disease relapse by Investigator determination, study-end or lost to follow-up, or death due to any cause. Due to the Covid-19 crisis causing significant delay of recruitment and the fact that we needed much more patients to identify patients with FGFR3 alterations, the study recruitment was prematurely stopped in November 2021 when 46 patients were screened and only 4 among 42 tested (9.5%) patients were identified with FGFR3 alterations. Two of the FGFR3 positive patients started treatment and the others were ineligible for the study. Since patients withdrawing from the study before completing the study period of 2 years cannot be included in the calculation of the 2-year RFS rate, the outcome results through premature study-end are presented.
Time Frame: Mean Relapse-free survival rate from start of treatment through premature study-end with a maximal follow-up of 62 weeks.
Population: 2 patients started treatment with Pemigatinib and were followed-up according to protocol through premature study-end.
Measure: Mean (Full Range); unit: weeks
Groups:
- Mean RFS for Patients Treated With Pemigatinib.: Mean RFS for patients treated with Pemigatinib and followed through premature study-end with a maximal follow up of 62 weeks.
Arm/Group | Mean RFS for Patients Treated With Pemigatinib.
Number analyzed (Participants) | 2
weeks | 26.6 [6.9 to 46.4]

2. Secondary Outcome: Mean Overall Survival After Start of Treatment With Pemigatinib.
Description: Mean Overall Survival of patients who started treatment with Pemigatinib is defined as the time from the start of treatment until the last date known alive, or death due to any cause through premature study-end.
Time Frame: Mean Overall Sturvival from start of treatment through premature study-end with a maximal follow-up of 62 weeks.
Population: 2 patients started treatment with Pemigatinib and were followed-up according to protocol through premature study-end with a maximal follow-up of 62 weeks.
Measure: Mean (Full Range); unit: weeks
Groups:
- Mean Overall Survival of Patients Treated With Pemigatinib.: Mean Overall Survival of patients who started treatment with Pemigatinib is defined as the time from the start of treatment until termination of the study or lost to follow-up, or death due to any cause through premature study-end.
Arm/Group | Mean Overall Survival of Patients Treated With Pemigatinib.
Number analyzed (Participants) | 2
weeks | 34.2 [6.9 to 61.6]

ADVERSE EVENTS:
Time Frame: From start of treatment to premature study end with a maximal follow-up of 62 weeks.
Arm/Group | Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=2)
high level of urea in blood (Blood and lymphatic system disorders) | 1 (1) — Grade 2
worsening visual acuity (Eye disorders) | 1 (1) — Grade 2
photophobia (Eye disorders) | 1 (1) — Grade 2
dygeusia (General disorders) | 1 (1) — Grade 3
weight loss (General disorders) | 1 (1) — Grade 2
hypotension (General disorders) | 1 (1) — Grade 2
xerostomia (General disorders) | 1 (1) — Grade 2
mouth ulcers (Infections and infestations) | 1 (1) — Grade 2
aching sole of foot (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 2
redness of basalioma (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 2
hairloss (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 2
xerosis cutis (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 2
mucositis mouth (Infections and infestations) | 1 (1) — Grade 2
fatique (General disorders) | 1 (1) — Grade 2

LIMITATIONS AND CAVEATS:
In 2020, we started in 5 Italian centers. We expected that 30% of the screened patients (pts) had FGFR3 alterations (F3). Due to the Covid-19 crisis (recruitment delay) and the fact that we needed more pts to identify F3, recruitment prematurely stopped in Nov. 2021 with 42 pts screened and only 4/42 tested identified with F3 (9%). Two out of 4 pts were ineligible and only 2 started treatment and were followed until Study-End in Nov. 2022 resulting in a limited follow-up of maximal 62 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT04294277/Prot_SAP_000.pdf